CLINICAL TRIAL: NCT03115177
Title: Can Addition of Doxycycline Perioperatively Reduce Propionibacterium Acnes in Shoulder Arthroplasty?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Allison Rao, Orthopaedic Surgery Resident, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15052002
Record Dates: First submitted 2016-04-25; First posted 2017-04-14 (Actual); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Doxycycline; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefazolin (Active Comparator): All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The control group will not receive any further antibiotic treatment.
  Interventions: Drug: Cefazolin
- Doxycycline+Cefazolin Group (Active Comparator): All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision.
  Interventions: Drug: Doxycycline; Drug: Cefazolin

INTERVENTIONS:
Drug: Doxycycline — The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision for total shoulder arthroplasty.
  Arms: Doxycycline+Cefazolin Group
Drug: Cefazolin

SUMMARY:
The purpose of this study is to investigate antibiotic treatment to target bacteria about the shoulder. This bacteria, Propionibacterium acnes, is detected in many revision shoulder surgeries and is thought to contribute to periprosthetic joint infections, pain, and failure of total shoulder arthroplasty as well as other shoulder surgeries. This study is investigating adding an FDA approved antibiotic that is commonly used for treatment of this bacteria and many common infections. The investigators will take intraoperative cultures to look for the presence or absence of specific bacteria. The investigators are conducting this trial to see if adding another antibiotic to specifically target this common bacteria found around the shoulder will be effective.

DETAILED DESCRIPTION:
Patients undergoing total and reverse shoulder arthroplasty for primary glenohumeral arthritis will be invited to participate in this study if patients meet inclusion and exclusion criteria. Patients will be randomized to receive either standard perioperative antibiotics with cefazolin or to the treatment group to receive doxycycline in addition to cefazolin. Patients will then undergo routine surgical treatment. 3 cultures from the superficial tissue, dermis, and glenohumeral joint will be taken and cultured for 14 days to detect any bacterial growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total shoulder arthroplasty at Rush University Medical Center

Exclusion Criteria:

* Patients with prior shoulder surgery of any kind
* Patients with a known infection or history of infection with clinical signs such as elevated erythrocyte sedimentation rate, C-reactive protein, positive culture aspiration
* Patients with a known allergy to doxycycline
* Patients with a known allergy to cefazolin or penicillin

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Rao, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefazolin: All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The control group will not receive any further antibiotic treatment.
  Cefazolin
- Cefazolin and Doxycycline: All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision.
  Doxycycline: The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision for total shoulder arthroplasty.
  Cefazolin
Period: Overall Study
Arm/Group | Cefazolin | Cefazolin and Doxycycline
Started | 27 | 29
Completed | 27 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Doxycycline+Cefazolin Group: All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision.
  Doxycycline: The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision for total shoulder arthroplasty.
  Cefazolin
- Total: Total of all reporting groups
Arm/Group | Cefazolin | Doxycycline+Cefazolin Group | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 16
  >=65 years | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8) | 67 (8) | 68 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 22 | 27 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (6) | 30 (6) | 30 (6)

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Culture
Description: Intraoperative cultures will be taken from all study participants and tested for detection of bacteria. These cultures were held for 14 days and tested for aerobic and anaerobic bacteria. Reported data are presented for the number of participants with a positive bacteria culture from the intraoperative samples.
Time Frame: 2 weeks
Measure: Number; unit: # Participants with Bacteria in Culture
Arm/Group | Cefazolin | Cefazolin and Doxycycline
Number analyzed (Participants) | 27 | 29
# Participants with Bacteria in Culture | 14 | 15

ADVERSE EVENTS:
Time Frame: Adverse events are recorded over the 1 year time period in which patients were recruited and participated in this study.
Groups:
- Control: All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The control group will not receive any further antibiotic treatment.
  Cefazolin
- Treatment: All patients will receive standard perioperative antibiotics with 2g of cefazolin within 1 hour of incision. The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision.
  Doxycycline: The treatment group will receive 100mg of doxycycline IV in addition to cefazolin within 1 hour of incision for total shoulder arthroplasty.
  Cefazolin
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT03115177/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT03115177/SAP_001.pdf